CLINICAL TRIAL: NCT02698410
Title: Efficacy and Safety of Lanreotide ATG 120 mg in Combination With Temozolomide in Subjects With Progressive Well Differentiated Thoracic Neuroendocrine Tumors. A Phase II, Multicentre, Single Arm, Open-label Trial.
Brief Title: Efficacy and Safety of Lanreotide Autogel (ATG) in Combination With Temozolomide in Subjects With Thoracic Neuroendocrine Tumors.
Acronym: ATLANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-93-52030-325; 2014-005579-10 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-03 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Neuroendocrine Tumours
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lanreotide; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lanreotide (Autogel formulation) and Temozolomide (Experimental): Lanreotide ATG 120 mg every 28 days, deep subcutaneous injection for a maximum of 48 weeks, for a total number of 12 injections.
  Temozolomide 250 mg hard capsules, for 5 consecutive days every 28 days, oral route, for a maximum of 48 weeks.
  Interventions: Drug: Lanreotide (Autogel formulation) and Temozolomide

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation) and Temozolomide

SUMMARY:
The purpose of the protocol is to evaluate the efficacy and safety of Lanreotide ATG 120 mg in combination with Temozolomide in subjects with unresectable advanced neuroendocrine tumours of the lung or thymus as Disease Control Rate at 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented unresectable advanced (locally or metastatic) well or moderately differentiated neuroendocrine tumors of the lung or thymus (typical and atypical carcinoids according to the World Health Organisation (WHO) 2004 criteria);
* Imaging documented progression within 12 months before screening visit (V1), according to RECIST criteria v 1.1;
* Measurable disease, as defined by RECIST criteria v 1.1, on a CT scan performed at screening visit (V1);
* Octreoscan or Ga68-DOTA-TATE/TOC/NOC-PET-TC within 12 months before screening visit (V1);
* Adequate liver, renal and bone marrow function.

Exclusion Criteria:

* Poorly differentiated neuroendocrine carcinoma and mixed Neuroendocrine tumours (NET), according to WHO 2004 criteria
* Neuroendocrine tumours other than lung or thymus
* Non-neuroendocrine thymic neoplasm
* Received a prior therapy with Peptide Receptor Radionuclide Therapy (PRRT) within 6 months prior to screening visit (V1)
* Treated with systemic therapies (chemotherapy, interferon-alpha, somatostatin analogues, molecular target therapies) within 1 month prior to screening visit (V1)
* Treated with a number of systemic therapy lines > 3 prior to screening visit (V1), and any of the following:

  1. for chemotherapy no more than 1 line prior to V1
  2. for somatostatin analogue no more than 1 line therapy, considered as treatment lasting more than 6 months, prior to V1 no therapy with Temozolomide (TMZ) prior to V1
  3. Received a prior therapy with Peptide Receptor Radionuclide Therapy (PRRT) within 6 months prior to screening visit (V1)
* Received external palliative radiotherapy within the last 28 days prior to screening visit (V1)
* Received locoregional therapies (Transarterial embolization, Transcatheter arterial chemoembolization, thermo-ablation with radio-frequency) and Selective internal radiotherapy within 3 months prior to screening visit (V1)
* Presence of symptomatic brain metastasis
* Subjects with symptomatic cholelithiasis at screening visit (V1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2019-02-08 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- Italy (10):
  - Oncologia Medica - Istituto Oncologico del Mediterraneo - IOM, Viagrande, Catania
  - Unità Operativa di Oncologia Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) S.r.l., IRCCS, Meldola
  - Unità Oncologia Medica Gastrointestinale e Tumori Neuroendocrini Istituto Europeo di Oncologia, IEO, Milan
  - Dipartimento di Endocrinologia e Oncologia Molecolare e Clinica , Università degli Studi, Napoli
  - Dipartimento di Oncologia Università di Torino Ospedale San Luigi Gonzaga, Orbassano
  - S.C di Oncologia Medica, Azienda Ospedaliera Universitaria di Perugia, Perugia
  - U.O. Oncologia - Azienda Ospedaliero-Universitaria Pisana Ospedale S. Chiara, Pisa
  - Oncologia Medica - Istituto Tumori Regina Elena San Gallicano, Roma
  - OUC di Oncologia- Azienda Ospedaliera Universitaria Integrata - Ospedale Borgo Roma, Verona

REFERENCES:
- [Derived] Ferolla P, Berruti A, Spada F, Brizzi MP, Ibrahim T, Marconcini R, Giuffrida D, Amoroso V, La Salvia A, Vaccaro V, Faggiano A, Colao A, Volante M, Ghizzoni S, Mazzanti P, Houchard A, Fazio N. Efficacy and Safety of Lanreotide Autogel and Temozolomide Combination Therapy in Progressive Thoracic Neuroendocrine Tumors (Carcinoid): Results from the Phase 2 ATLANT Study. Neuroendocrinology. 2023;113(3):332-342. doi: 10.1159/000526811. Epub 2022 Aug 31. PMID 36044870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This pilot study was conducted at 11 investigational sites in Italy between 06 July 2016 and 18 June 2019.
Pre-assignment Details: The study consisted of a screening period (maximum 4 weeks), followed by an open label treatment period of up to a maximum of 52 weeks or until disease progression, death or unacceptable toxicity, or subject/physician decision.
Groups:
- Lanreotide Autogel (ATG) Plus Temozolomide: Lanreotide ATG 120 milligrams (mg) was administered by deep subcutaneous injection on Day 1 (baseline) and every 28 days for up to 52 weeks. Participants also received temozolomide 250 mg capsule orally once daily for 5 consecutive days every 28 days for up to 52 weeks. The dose of temozolomide could subsequently be reduced to 180 mg daily for 5 consecutive days every 28 days in case of bone marrow toxicity.
Period: Overall Study
Arm/Group | Lanreotide Autogel (ATG) Plus Temozolomide
Started | 40
Completed | 36
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The Intention-to-treat (ITT)/Safety population included all participants who received at least 1 dose of study medication (either lanreotide ATG 120 mg or temozolomide).
Groups:
- Lanreotide ATG Plus Temozolomide: Lanreotide ATG 120 mg was administered by deep subcutaneous injection on Day 1 (baseline) and every 28 days for up to 52 weeks. Participants also received temozolomide 250 mg capsule orally once daily for 5 consecutive days every 28 days for up to 52 weeks. The dose of temozolomide could subsequently be reduced to 180 mg daily for 5 consecutive days every 28 days in case of bone marrow toxicity.
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) Assessed Locally at Month 9
Description: Responders were participants who showed disease control according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria v 1.1 assessed locally by the investigator. The DCR was defined as complete response (CR), partial response (PR) or stable disease (SD) according to RECIST criteria v1.1. A sensitivity analysis-1 of local DCR was performed excluding participants withdrawn before 9 months with reason other than progressive disease (PD) or missing assessment and considering participants with PD prior or at 9 months as failures. In addition, a sensitivity analysis-2 was performed in order to consider assessments done between 7.5 and 10.5 months as 9 months assessments when 9-month assessment was missing using same methodology, i.e. considering PD prior or at 9 months and participants withdrawn with other or missing reasons as failures.
Time Frame: Up to Month 9; for sensitivity analysis-2, up to 10.5 months
Population: The ITT/Safety population included all participants who received at least 1 dose of study medication (either lanreotide ATG 120 mg or temozolomide).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
percentage of participants
  DCR at Month 9 | 35.0 [20.63 to 51.68]
  Sensitivity analysis-1: number analyzed (Participants) | 31
  Sensitivity analysis-1 | 45.2 [27.32 to 63.97]
  Sensitivity analysis-2 | 45.0 [29.26 to 61.51]
Statistical Analysis 1: Comparison: Lanreotide ATG Plus Temozolomide; Comparison of DCR to 30% clinically relevant threshold; Test type: Other; p = 0.2968, Binomial proportion test — One-sided p-value estimated using an exact binomial proportion test for one-way tables comparing DCR to 30%
Statistical Analysis 2: Comparison: Lanreotide ATG Plus Temozolomide; Comparison of DCR to 10% clinically relevant threshold; Test type: Other; p < 0.0001, Binomial proportion test — One-sided p-value estimated using an exact binomial proportion test for one-way tables comparing DCR to 10%
Statistical Analysis 3: Comparison: Lanreotide ATG Plus Temozolomide; Sensitivity Analyisis-1: Comparison of DCR to 30% clinically relevant threshold; Test type: Other; p = 0.0534, Binomial proportion test — One-sided p-value estimated using an exact binomial proportion test for one-way tables comparing DCR to 30%
Statistical Analysis 4: Comparison: Lanreotide ATG Plus Temozolomide; Sensitivity Analyisis-1: Comparison of DCR to 10% clinically relevant threshold; Test type: Other; p < 0.0001, Binomial proportion test — One-sided p-value estimated using an exact binomial proportion test for one-way tables comparing DCR to 10%
Statistical Analysis 5: Comparison: Lanreotide ATG Plus Temozolomide; Sensitivity Analyisis-2: Comparison of DCR to 30% clinically relevant threshold; Test type: Other; p = 0.032, Binomial proportion test — One-sided p-value estimated using an exact binomial proportion test for one-way tables comparing DCR to 30%
Statistical Analysis 6: Comparison: Lanreotide ATG Plus Temozolomide; Sensitivity Analyisis-2: Comparison of DCR to 10% clinically relevant threshold; Test type: Other; p < 0.0001, Binomial proportion test — One-sided p-value estimated using an exact binomial proportion test for one-way tables comparing DCR to 10%

2. Secondary Outcome: DCR Assessed Centrally at Month 9
Description: The DCR was defined as SD, PR or CR according to RECIST criteria v1.1. A second set of the original computed tomography (CT) scan images were used for a centralized RECIST v1.1 assessment by an independent radiologist.
Time Frame: Up to Month 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
percentage of participants | 28.2 [15.00 to 44.87]

3. Secondary Outcome: Median Progression Free Survival (PFS) Assessed Locally and Centrally
Description: The PFS was defined as the time from the first treatment administration to disease progression according to RECIST criteria v 1.1 or death from any cause. The PFS was assessed locally by the investigator and centrally by an independent radiologist. The distribution of PFS times was estimated using the Kaplan-Meier method. The PFS of participants who were lost to follow-up and those who had not progressed at end of study were censored at the date of the last disease assessment.
Time Frame: From Day 1 up to end of study, 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
weeks
  Local assessment | 37.1 [24.1 to 52.9]
  Central assessment | 37.1 [24.1 to 56.0]

4. Secondary Outcome: Median Time to Response (TTR) Assessed Locally and Centrally
Description: The TTR was defined as the time from first treatment administration to the first objective tumor response (PR or CR according to RECIST criteria v 1.1). The TTR was assessed locally by the investigator and centrally by an independent radiologist. The distribution of TTR was estimated using the Kaplan-Meier method. The TTR of participants who were lost to follow-up or died prior to any objective tumor response were censored at the date of the last disease assessment.
Time Frame: From Day 1 up to end of study, 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
weeks
  Local assessment | NA [NA to NA] — Not computed as the median TTR could not be estimated due to the low number of participants with an objective response (OR).
  Central assessment | NA [NA to NA] — Not computed as the median TTR could not be estimated due to the low number of participants with an OR.

5. Secondary Outcome: Median Duration of Response (DOR) Assessed Locally and Centrally
Description: The DOR was defined as the time from onset of the first objective tumor response (PR or CR) to objective tumor progression (PD) according to RECIST criteria v 1.1. The DOR was assessed locally by the investigator and centrally by an independent radiologist.
Time Frame: From Day 1 up to end of study, 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
weeks
  Local assessment | NA [NA to NA] — The median DOR could not be estimated due to the low number of participants with an OR with no documented PD.
  Central assessment | NA [NA to NA] — The median DOR could not be estimated due to the low number of participants with an OR with no documented PD.

6. Secondary Outcome: Median Time to Progression (TTP) Assessed Locally and Centrally
Description: The TTP was defined as the time from first treatment administration to the first objective tumor progression (PD) according to RECIST criteria v 1.1. The TTP was assessed locally by the investigator and centrally by an independent radiologist. The distribution of TTP times was estimated using the Kaplan-Meier method. The TTP of participants who were lost to follow-up, and those who had not progressed at end of study were censored at the date of the last disease assessment.
Time Frame: From Day 1 up to end of study, 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
weeks
  Local assessment | 37.1 [26.4 to 55.1]
  Central assessment | 37.1 [24.1 to 56.0]

7. Secondary Outcome: Best Overall Response (BOR) Assessed Locally and Centrally
Description: The BOR was defined as the highest OR achieved by the participant from the time of first treatment until disease progression/recurrence or the end of study according to RECIST criteria v1.1 and was classified as: CR > PR > Non-CR/Non-progressive disease (NCR/NPD) > SD > PD > ND > not evaluable (NE). The BOR was assessed locally by the investigator and centrally by an independent radiologist. Percentages are based on the number of participants in the ITT/Safety population with non-missing observations.
Time Frame: From Day 1 up to end of study, 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 39
percentage of participants
  Local assessment: CR | 0
  Local assessment: PR | 7.7
  Local assessment: SD | 71.8
  Local assessment: NCR/NPD | 0
  Local assessment: PD | 20.5
  Local assessment: NE | 0
  Local assessment: Not applicable | 0
  Central assessment: CR: number analyzed (Participants) | 38
  Central assessment: CR | 0
  Central assessment: PR: number analyzed (Participants) | 38
  Central assessment: PR | 13.2
  Central assessment: SD: number analyzed (Participants) | 38
  Central assessment: SD | 65.8
  Central assessment: NCR/NPD: number analyzed (Participants) | 38
  Central assessment: NCR/NPD | 2.6
  Central assessment: PD: number analyzed (Participants) | 38
  Central assessment: PD | 15.8
  Central assessment: NE: number analyzed (Participants) | 38
  Central assessment: NE | 0
  Central assessment: Not applicable: number analyzed (Participants) | 38
  Central assessment: Not applicable | 2.6

8. Secondary Outcome: Objective Response Rate (ORR) Assessed Locally and Centrally at Months 9 and 12
Description: The ORR was defined as the percentage of participants with CR or PR according to RECIST criteria v1.1. The ORR was assessed locally by the investigator and centrally by an independent radiologist. The ORR was based on the participants with PD prior to 9 and 12 months with respectively PD at 9 and 12 months, and participants withdrawn before the assessment for reason other than PD or missing as failures.
Time Frame: Months 9 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
percentage of participants
  Local assessment: Month 9 | 2.5 [0.06 to 13.16]
  Local assessment: Month 12 | 2.5 [0.06 to 13.16]
  Central assessment: Month 9 | 5.1 [0.63 to 17.32]
  Central assessment: Month 12 | 2.6 [0.06 to 13.48]

9. Secondary Outcome: DCR Assessed Locally and Centrally at Month 12
Description: The DCR was defined as SD, PR or CR according to RECIST criteria v1.1. The DCR was assessed locally by the investigator and centrally by an independent radiologist.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
percentage of participants
  Local assessment | 17.5 [7.34 to 32.78]
  Central assessment | 15.4 [5.86 to 30.53]

10. Secondary Outcome: DCR Assessed Locally and Centrally at Month 9 by Carcinoid Type
Description: The influence of type of carcinoid [typical, atypical and undetermined carcinoid neuroendocrine tumors (NET)] on the local and central DCR at 9 months was analysed. Typical carcinoids were defined with absent foci of necrosis and mitotic count < 2 mitoses/2 millimeters^2 (mm^2); atypical carcinoids were defined with presence of foci of necrosis and/or 2 mitoses/2 mm^2 <= mitotic count <= 10 mitoses/2 mm^2; and carcinoid NET were defined as confirmed carcinoid without foci of necrosis and/or mitotic count reported. The DCR was assessed locally by the investigator and centrally by an independent radiologist.
Time Frame: Up to Month 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
percentage of participants
  Local assessment: Typical carcinoid: number analyzed (Participants) | 8
  Local assessment: Typical carcinoid | 12.5 [0.32 to 52.65]
  Local assessment: Atypical carcinoid: number analyzed (Participants) | 21
  Local assessment: Atypical carcinoid | 47.6 [25.71 to 70.22]
  Local assessment: Carcinoid NET: number analyzed (Participants) | 11
  Local assessment: Carcinoid NET | 27.3 [6.02 to 60.97]
  Central assessment: Typical carcinoid: number analyzed (Participants) | 8
  Central assessment: Typical carcinoid | 0 [NA to NA] — The confidence interval could not be calculated due to no events.
  Central assessment: Atypical carcinoid: number analyzed (Participants) | 21
  Central assessment: Atypical carcinoid | 35.0 [15.39 to 59.22]
  Central assessment: Carcinoid NET: number analyzed (Participants) | 11
  Central assessment: Carcinoid NET | 36.4 [10.93 to 69.21]

11. Secondary Outcome: Percentage of Biochemical Responders According to Chromogranin A (CgA) Plasma Levels
Description: Participants with baseline CgA plasma levels greater than the upper limit of normal (ULN) were assessed for a biochemical response. A biochemical responder was defined as a participant who had a decrease of CgA >= 50% compared to baseline, while biochemical SD was defined as a decrease < 50% or an increase <= 25% compared to baseline. Biochemical non-responders had an increase >25% compared to baseline. Baseline was defined as value at Day 1.
Time Frame: Baseline (Day 1) and Week 4, 12, 24, 36 and 52
Population: The ITT/Safety population included all participants who received at least 1 dose of study medication (either lanreotide ATG 120 mg or temozolomide). Only participants with baseline CgA levels greater than ULN were analysed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 24
percentage of participants
  Week 4: Responders: number analyzed (Participants) | 22
  Week 4: Responders | 27.3 [9.36 to 45.13]
  Week 4: SD: number analyzed (Participants) | 22
  Week 4: SD | 59.1 [31.31 to 72.2]
  Week 4: Non-responders: number analyzed (Participants) | 22
  Week 4: Non-responders | 13.6 [2.55 to 31.22]
  Week 12: Responders: number analyzed (Participants) | 16
  Week 12: Responders | 37.5 [11.89 to 54.28]
  Week 12: SD: number analyzed (Participants) | 16
  Week 12: SD | 37.5 [11.89 to 54.28]
  Week 12: Non-responders: number analyzed (Participants) | 16
  Week 12: Non-responders | 25.0 [5.73 to 43.66]
  Week 24: Responders: number analyzed (Participants) | 13
  Week 24: Responders | 23.1 [5.04 to 53.81]
  Week 24: SD: number analyzed (Participants) | 13
  Week 24: SD | 30.8 [9.09 to 61.43]
  Week 24: Non-responders: number analyzed (Participants) | 13
  Week 24: Non-responders | 46.2 [19.22 to 74.87]
  Week 36: Responders: number analyzed (Participants) | 11
  Week 36: Responders | 36.4 [9.09 to 61.43]
  Week 36: SD: number analyzed (Participants) | 11
  Week 36: SD | 27.3 [5.04 to 53.81]
  Week 36: Non-responders: number analyzed (Participants) | 11
  Week 36: Non-responders | 36.4 [9.09 to 61.43]
  Week 52: Responders: number analyzed (Participants) | 8
  Week 52: Responders | 12.5 [0.28 to 48.25]
  Week 52: SD: number analyzed (Participants) | 8
  Week 52: SD | 50.0 [13.7 to 78.8]
  Week 52: Non-responders: number analyzed (Participants) | 8
  Week 52: Non-responders | 37.5 [7.49 to 70.07]

12. Secondary Outcome: Neuron-Specific Enolase (NSE) and CgA Biomarker Levels
Description: The NSE and CgA levels were classified according to ULN as follows: < 1 ULN, 1-2 ULN and > 2 ULN. Baseline was defined as value at Day 1. Percentages are based on the number of participants in the ITT/Safety population who attended the visit with non-missing observations.
Time Frame: Baseline and Weeks 4, 12, 24, 36 and 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
percentage of participants
  CgA: Baseline: <1 ULN | 40.0
  CgA: Baseline: 1-2 ULN | 15.0
  CgA: Baseline: >2 ULN | 45.0
  CgA: Week 4: <1 ULN: number analyzed (Participants) | 35
  CgA: Week 4: <1 ULN | 34.3
  CgA: Week 4: 1-2 ULN: number analyzed (Participants) | 35
  CgA: Week 4: 1-2 ULN | 22.9
  CgA: Week 4: >2 ULN: number analyzed (Participants) | 35
  CgA: Week 4: >2 ULN | 42.9
  CgA: Week 12: <1 ULN: number analyzed (Participants) | 28
  CgA: Week 12: <1 ULN | 46.4
  CgA: Week 12: 1-2 ULN: number analyzed (Participants) | 28
  CgA: Week 12: 1-2 ULN | 17.9
  CgA: Week 12: >2 ULN: number analyzed (Participants) | 28
  CgA: Week 12: >2 ULN | 35.7
  CgA: Week 24: <1 ULN: number analyzed (Participants) | 20
  CgA: Week 24: <1 ULN | 30.0
  CgA: Week 24: 1-2 ULN: number analyzed (Participants) | 20
  CgA: Week 24: 1-2 ULN | 25.0
  CgA: Week 24: >2 ULN: number analyzed (Participants) | 20
  CgA: Week 24: >2 ULN | 45.0
  CgA: Week 36: <1 ULN: number analyzed (Participants) | 16
  CgA: Week 36: <1 ULN | 31.3
  CgA: Week 36: 1-2 ULN: number analyzed (Participants) | 16
  CgA: Week 36: 1-2 ULN | 12.5
  CgA: Week 36: >2 ULN: number analyzed (Participants) | 16
  CgA: Week 36: >2 ULN | 56.3
  CgA: Week 52: <1 ULN: number analyzed (Participants) | 11
  CgA: Week 52: <1 ULN | 27.3
  CgA: Week 52: 1-2 ULN: number analyzed (Participants) | 11
  CgA: Week 52: 1-2 ULN | 9.1
  CgA: Week 52: >2 ULN: number analyzed (Participants) | 11
  CgA: Week 52: >2 ULN | 63.6
  NSE: Baseline: <1 ULN | 65.0
  NSE: Baseline: 1-2 ULN | 25.0
  NSE: Baseline: >2 ULN | 10.0
  NSE: Week 4: <1 ULN: number analyzed (Participants) | 35
  NSE: Week 4: <1 ULN | 62.9
  NSE: Week 4: 1-2 ULN: number analyzed (Participants) | 35
  NSE: Week 4: 1-2 ULN | 25.7
  NSE: Week 4: >2 ULN: number analyzed (Participants) | 35
  NSE: Week 4: >2 ULN | 11.4
  NSE: Week 12: <1 ULN: number analyzed (Participants) | 28
  NSE: Week 12: <1 ULN | 78.6
  NSE: Week 12: 1-2 ULN: number analyzed (Participants) | 28
  NSE: Week 12: 1-2 ULN | 17.9
  NSE: Week 12: >2 ULN: number analyzed (Participants) | 28
  NSE: Week 12: >2 ULN | 3.6
  NSE: Week 24: <1 ULN: number analyzed (Participants) | 20
  NSE: Week 24: <1 ULN | 80.0
  NSE: Week 24: 1-2 ULN: number analyzed (Participants) | 20
  NSE: Week 24: 1-2 ULN | 10.0
  NSE: Week 24: >2 ULN: number analyzed (Participants) | 20
  NSE: Week 24: >2 ULN | 10.0
  NSE: Week 36: <1 ULN: number analyzed (Participants) | 16
  NSE: Week 36: <1 ULN | 87.5
  NSE: Week 36: 1-2 ULN: number analyzed (Participants) | 16
  NSE: Week 36: 1-2 ULN | 6.3
  NSE: Week 36: >2 ULN: number analyzed (Participants) | 16
  NSE: Week 36: >2 ULN | 6.3
  NSE: Week 52: <1 ULN: number analyzed (Participants) | 11
  NSE: Week 52: <1 ULN | 63.6
  NSE: Week 52: 1-2 ULN: number analyzed (Participants) | 11
  NSE: Week 52: 1-2 ULN | 18.2
  NSE: Week 52: >2 ULN: number analyzed (Participants) | 11
  NSE: Week 52: >2 ULN | 18.2

13. Secondary Outcome: Influence of Biomarkers Expression on Locally and Centrally Assessed PFS
Description: The following biomarkers were investigated: Immunohistochemistry assay human somatostatin receptors 2 (SSTR2) including human epidermal growth factor receptor 2 (HER-2) score [0, 1+, 2+, 3+ and positive (+ve) versus negative (-ve)]; hormone receptor score (H-score) (from 0 to 300 as quantitative variable and +ve versus -ve); immunoreactive score (IRS) score (from 0 to 12 and reference for hazard ratio was 0-1). Ki67 index (from 0% to 100% and reference for hazard ratio was 4%-25%). O^6-methylguanine-DNA methyltransferase (MGMT) expression including percentage of +ve nuclei stained and methylated sites and H-score (from 0 to 300 as quantitative variable). For all these categories, higher score indicates a higher expression of biomarkers. Carcinoid type (typical or NET) was also investigated. Prognostic value of biomarkers expression at screening on PFS were assessed locally and centrally using univariate cox proportional hazard models.
Time Frame: From Screening period (-4 weeks) up to Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
hazard ratio
  Local: SSTR2: HER-2 score; +ve (2+, 3+): number analyzed (Participants) | 26
  Local: SSTR2: HER-2 score; +ve (2+, 3+) | 0.71 [0.26 to 1.92]
  Local: SSTR2: H-score; +ve (>= 50): number analyzed (Participants) | 26
  Local: SSTR2: H-score; +ve (>= 50) | 0.66 [0.25 to 1.71]
  Local: SSTR2: IRS score; 2-3: number analyzed (Participants) | 26
  Local: SSTR2: IRS score; 2-3 | 0.31 [0.04 to 2.61]
  Local: SSTR2: IRS score; 4-8: number analyzed (Participants) | 26
  Local: SSTR2: IRS score; 4-8 | 0.90 [0.31 to 2.61]
  Local: SSTR2: IRS score; 9-12: number analyzed (Participants) | 26
  Local: SSTR2: IRS score; 9-12 | 0.12 [0.01 to 0.99]
  Local: Ki67: <4: number analyzed (Participants) | 20
  Local: Ki67: <4 | 1.08 [0.13 to 8.93]
  Local: Ki67: >=25: number analyzed (Participants) | 20
  Local: Ki67: >=25 | 1.68 [0.37 to 7.70]
  Local: MGMT: +ve nuclei stained; +ve (>=5%): number analyzed (Participants) | 26
  Local: MGMT: +ve nuclei stained; +ve (>=5%) | 2.06 [0.27 to 15.69]
  Local: MGMT: Methylated sites; +ve (>10%): number analyzed (Participants) | 24
  Local: MGMT: Methylated sites; +ve (>10%) | 0.41 [0.05 to 3.20]
  Local: MGMT: H-score: number analyzed (Participants) | 26
  Local: MGMT: H-score | 1.00 [1.00 to 1.01]
  Local: Carcinoid type: Typical | 1.05 [0.36 to 3.07]
  Local: Carcinoid type: Carcinoid NET | 1.59 [0.64 to 3.93]
  Central: SSTR2: HER-2 score; +ve (2+, 3+): number analyzed (Participants) | 26
  Central: SSTR2: HER-2 score; +ve (2+, 3+) | 0.50 [0.18 to 1.39]
  Central: SSTR2: H-score; +ve (>= 50): number analyzed (Participants) | 26
  Central: SSTR2: H-score; +ve (>= 50) | 0.36 [0.12 to 1.04]
  Central: SSTR2: IRS score; 2-3: number analyzed (Participants) | 26
  Central: SSTR2: IRS score; 2-3 | 0.78 [0.16 to 3.92]
  Central: SSTR2: IRS score; 4-8: number analyzed (Participants) | 26
  Central: SSTR2: IRS score; 4-8 | 0.88 [0.28 to 2.76]
  Central: SSTR2: IRS score; 9-12: number analyzed (Participants) | 26
  Central: SSTR2: IRS score; 9-12 | 0.10 [0.01 to 0.89]
  Central: Ki67: <4: number analyzed (Participants) | 20
  Central: Ki67: <4 | 0.00 [0.00 to NA] — The 95% confidence interval upper bound not computed due to low number of participants in the given category with an event.
  Central: Ki67: >=25: number analyzed (Participants) | 20
  Central: Ki67: >=25 | 2.75 [0.55 to 13.76]
  Central: MGMT: +ve nuclei stained; +ve (>=5%): number analyzed (Participants) | 26
  Central: MGMT: +ve nuclei stained; +ve (>=5%) | 2.11 [0.27 to 16.34]
  Central: MGMT: Methylated sites; +ve (>10%): number analyzed (Participants) | 24
  Central: MGMT: Methylated sites; +ve (>10%) | 0.73 [0.16 to 3.33]
  Central: MGMT: H-score: number analyzed (Participants) | 26
  Central: MGMT: H-score | 1.00 [0.99 to 1.01]
  Central: Carcinoid type: Typical | 0.99 [0.35 to 2.82]
  Central: Carcinoid type: Carcinoid NET | 0.61 [0.20 to 1.89]

14. Secondary Outcome: Influence of Biomarkers Expression on Locally and Centrally Assessed ORR at Months 9 and 12
Description: The following biomarkers were investigated: Immunohistochemistry assay SSTR2 including HER-2 score (0, 1+, 2+, 3+); H-score (from 0 to 300 as quantitative variable); IRS score (from 0 to 12). Ki67 index (from 0% to 100%). MGMT expression including percentage of +ve nuclei stained and methylated sites and H-score (from 0 to 300 as quantitative variable). For all these categories, higher score indicates a higher expression of biomarkers. Less than 5 OR (CR or PR) events were reported, therefore this analysis was not performed.
Time Frame: Screening period, Months 9 and 12
Population: No analysis on ORR at 9 and 12 months was performed due to insufficient number of participants with OR events.
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 0

15. Secondary Outcome: Influence of Biomarkers Expression on Locally and Centrally Assessed DCR at Months 9 and 12
Description: The following biomarkers were investigated: Immunohistochemistry assay SSTR2 including HER-2 score (0, 1+, 2+, 3+ and +ve versus -ve); H-score (from 0 to 300 as quantitative variable and +ve versus -ve); IRS score (from 0 to 12 and reference for odds ratio was 0-1). Ki67 index (from 0% to 100% and reference for odds ratio was 4%-25%). MGMT expression including percentage of +ve nuclei stained and methylated sites and H-score (from 0 to 300 as quantitative variable). For all these categories, higher score indicates a higher expression of biomarkers. Carcinoid type (typical or NET) was also investigated. Prognostic value of biomarkers expression at screening on DCR were assessed locally and centrally using univariate logistic regression models.
Time Frame: Screening period, Months 9 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
odds ratio
  Month 9: Local: SSTR2: HER-2 score; +ve (2+, 3+): number analyzed (Participants) | 26
  Month 9: Local: SSTR2: HER-2 score; +ve (2+, 3+) | 0.90 [0.18 to 4.55]
  Month 9: Local: SSTR2: H-score; +ve (>= 50): number analyzed (Participants) | 26
  Month 9: Local: SSTR2: H-score; +ve (>= 50) | 0.78 [0.16 to 3.79]
  Month 9: Local: SSTR2: IRS score; 2-3: number analyzed (Participants) | 26
  Month 9: Local: SSTR2: IRS score; 2-3 | NA [NA to NA] — Not calculated due to low number of participants in the given category with an event.
  Month 9: Local: SSTR2: IRS score; 4-8: number analyzed (Participants) | 26
  Month 9: Local: SSTR2: IRS score; 4-8 | 0.67 [0.07 to 6.11]
  Month 9: Local: SSTR2: IRS score; 9-12: number analyzed (Participants) | 26
  Month 9: Local: SSTR2: IRS score; 9-12 | 12.00 [0.80 to 180.97]
  Month 9: Local: Ki67: <4: number analyzed (Participants) | 20
  Month 9: Local: Ki67: <4 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 9: Local: Ki67: >=25: number analyzed (Participants) | 20
  Month 9: Local: Ki67: >=25 | 1.67 [0.09 to 31.87]
  Month 9:Local: MGMT: +ve nuclei stained; +ve(>=5%): number analyzed (Participants) | 26
  Month 9:Local: MGMT: +ve nuclei stained; +ve(>=5%) | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 9: Local: MGMT: Methylated sites; +ve (>10%): number analyzed (Participants) | 24
  Month 9: Local: MGMT: Methylated sites; +ve (>10%) | 3.25 [0.25 to 41.91]
  Month 9: Local: MGMT: H-score: number analyzed (Participants) | 26
  Month 9: Local: MGMT: H-score | 0.99 [0.98 to 1.00]
  Month 9: Local: Carcinoid type: Typical | 0.16 [0.02 to 1.51]
  Month 9: Local: Carcinoid type: Carcinoid NET | 0.41 [0.09 to 2.00]
  Month 9: Central: SSTR2: HER-2 score; +ve (2+, 3+): number analyzed (Participants) | 26
  Month 9: Central: SSTR2: HER-2 score; +ve (2+, 3+) | 1.40 [0.26 to 7.58]
  Month 9: Central: SSTR2: H-score; +ve (>= 50): number analyzed (Participants) | 26
  Month 9: Central: SSTR2: H-score; +ve (>= 50) | 2.25 [0.42 to 12.09]
  Month 9: Central: SSTR2: IRS score; 2-3: number analyzed (Participants) | 26
  Month 9: Central: SSTR2: IRS score; 2-3 | 3.00 [0.12 to 73.64]
  Month 9: Central: SSTR2: IRS score; 4-8: number analyzed (Participants) | 26
  Month 9: Central: SSTR2: IRS score; 4-8 | 0.67 [0.07 to 6.11]
  Month 9: Central: SSTR2: IRS score; 9-12: number analyzed (Participants) | 26
  Month 9: Central: SSTR2: IRS score; 9-12 | 12.00 [0.80 to 180.97]
  Month 9: Central: Ki67: <4: number analyzed (Participants) | 20
  Month 9: Central: Ki67: <4 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 9: Central: Ki67: >=25: number analyzed (Participants) | 20
  Month 9: Central: Ki67: >=25 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 9:Central:MGMT:+ve nuclei stained; +ve(>=5%): number analyzed (Participants) | 26
  Month 9:Central:MGMT:+ve nuclei stained; +ve(>=5%) | 0.50 [0.03 to 9.08]
  Month 9:Central: MGMT: Methylated sites; +ve(>10%): number analyzed (Participants) | 24
  Month 9:Central: MGMT: Methylated sites; +ve(>10%) | 5.00 [0.38 to 66.01]
  Month 9: Central: MGMT: H-score: number analyzed (Participants) | 26
  Month 9: Central: MGMT: H-score | 1.00 [0.99 to 1.01]
  Month 9: Central: Carcinoid type: Typical | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 9: Central: Carcinoid type: Carcinoid NET | 1.06 [0.23 to 4.92]
  Month 12: Local: SSTR2: HER-2 score; +ve (2+, 3+): number analyzed (Participants) | 26
  Month 12: Local: SSTR2: HER-2 score; +ve (2+, 3+) | 3.00 [0.28 to 31.63]
  Month 12: Local: SSTR2: H-score; +ve (>= 50): number analyzed (Participants) | 26
  Month 12: Local: SSTR2: H-score; +ve (>= 50) | 4.40 [0.42 to 46.24]
  Month 12: Local: SSTR2: IRS score; 2-3: number analyzed (Participants) | 26
  Month 12: Local: SSTR2: IRS score; 2-3 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 12: Local: SSTR2: IRS score; 4-8: number analyzed (Participants) | 26
  Month 12: Local: SSTR2: IRS score; 4-8 | 0.70 [0.04 to 13.18]
  Month 12: Local: SSTR2: IRS score; 9-12: number analyzed (Participants) | 26
  Month 12: Local: SSTR2: IRS score; 9-12 | 10.50 [0.67 to 165.11]
  Month 12: Local: Ki67: <4: number analyzed (Participants) | 20
  Month 12: Local: Ki67: <4 | NA [NA to NA] — Not calculated due to low number of participants in the given category with an event.
  Month 12: Local: Ki67: >=25: number analyzed (Participants) | 20
  Month 12: Local: Ki67: >=25 | NA [NA to NA] — Not calculated due to low number of participants in the given category with an event.
  Month 12:Local:MGMT: +ve nuclei stained; +ve(>=5%): number analyzed (Participants) | 26
  Month 12:Local:MGMT: +ve nuclei stained; +ve(>=5%) | 0.20 [0.01 to 3.91]
  Month 12: Local: MGMT: Methylated sites; +ve(>10%): number analyzed (Participants) | 24
  Month 12: Local: MGMT: Methylated sites; +ve(>10%) | 2.13 [0.15 to 29.66]
  Month 12: Local: MGMT: H-score: number analyzed (Participants) | 26
  Month 12: Local: MGMT: H-score | 0.99 [0.96 to 1.01]
  Month 12: Local: Carcinoid type: Typical | 0.46 [0.04 to 4.67]
  Month 12: Local: Carcinoid type: Carcinoid NET | 0.32 [0.03 to 3.15]
  Month 12: Central: SSTR2: HER-2 score; +ve(2+, 3+): number analyzed (Participants) | 26
  Month 12: Central: SSTR2: HER-2 score; +ve(2+, 3+) | 2.08 [0.19 to 23.30]
  Month 12: Central: SSTR2: H-score; +ve (>= 50): number analyzed (Participants) | 26
  Month 12: Central: SSTR2: H-score; +ve (>= 50) | 3.00 [0.27 to 33.49]
  Month 12: Central: SSTR2: IRS score; 2-3: number analyzed (Participants) | 26
  Month 12: Central: SSTR2: IRS score; 2-3 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 12: Central: SSTR2: IRS score; 4-8: number analyzed (Participants) | 26
  Month 12: Central: SSTR2: IRS score; 4-8 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 12: Central: SSTR2: IRS score; 9-12: number analyzed (Participants) | 26
  Month 12: Central: SSTR2: IRS score; 9-12 | 10.50 [0.67 to 165.11]
  Month 12: Central: Ki67: <4: number analyzed (Participants) | 20
  Month 12: Central: Ki67: <4 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 12: Central: Ki67: >=25: number analyzed (Participants) | 20
  Month 12: Central: Ki67: >=25 | NA [NA to NA] — The 95% confidence interval could not be computed as the odds ratio is <0.001.
  Month 12:Central:MGMT:+ve nuclei stained;+ve(>=5%): number analyzed (Participants) | 26
  Month 12:Central:MGMT:+ve nuclei stained;+ve(>=5%) | 0.14 [0.01 to 2.94]
  Month 12:Central: MGMT: Methylated sites;+ve(>10%): number analyzed (Participants) | 24
  Month 12:Central: MGMT: Methylated sites;+ve(>10%) | 3.00 [0.20 to 44.36]
  Month 12: Central: MGMT: H-score: number analyzed (Participants) | 26
  Month 12: Central: MGMT: H-score | 0.99 [0.96 to 1.01]
  Month 12: Central: Carcinoid type: Typical | 0.57 [0.05 to 6.08]
  Month 12: Central: Carcinoid type: Carcinoid NET | 0.40 [0.04 to 4.11]

16. Secondary Outcome: Coefficient of Agreement Between Central and Local Assessment of Tumor Radiological Response at Month 9
Description: Differences between central radiology review and local investigator review were assessed according to the DCR status and the number of agreements and disagreements between the evaluators (central versus local) along with the p-values from the kappa test. A kappa statistic was used to evaluate the concordance between the central and the local review.
Time Frame: Month 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: kappa coefficient
Arm/Group | Lanreotide ATG Plus Temozolomide
Number analyzed (Participants) | 40
kappa coefficient | 0.71 [0.48 to 0.94]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of the first treatment (Day 1) until 4 weeks after the end of the last study treatment, up to a maximum of 52 weeks.
Description: The ITT/Safety population included all participants who received at least 1 dose of study medication (either lanreotide ATG 120 mg or temozolomide). All-cause mortality occurred in both treatment period and follow-up period were reported.
Arm/Group | Lanreotide ATG Plus Temozolomide
All-Cause Mortality (participants affected / at risk) | 9/40
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide ATG Plus Temozolomide (N=40)
Death (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide ATG Plus Temozolomide (N=40)
Nausea (Gastrointestinal disorders) | 21 (42)
Vomiting (Gastrointestinal disorders) | 13 (24)
Diarrhoea (Gastrointestinal disorders) | 12 (36)
Constipation (Gastrointestinal disorders) | 8 (26)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 8 (8)
Pyrexia (General disorders) | 6 (6)
Pain (General disorders) | 4 (4)
Influenza like illness (General disorders) | 3 (3)
Fatigue (General disorders) | 2 (4)
Chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Weight decreased (Investigations) | 7 (7)
Blood cholesterol increased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 4 (7)
Blood creatinine increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 2 (2)
Blood triglycerides increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (5)
White blood cell count decreased (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Glucose tolerance decreased (Investigations) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Vitamin b12 decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Angular cheilitis (Infections and infestations) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 4 (5)
Sciatica (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (3)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results are owned by the Sponsor and data communication collected in a center by the investigator is allowed only after publication of aggregate results of the study by the Sponsor. If an investigator intends to communicate data, the Sponsor must be informed and should review the manuscript/publication before its submission. The investigator should accept any Sponsor comments provided they are not in contrast to the reliability of data, with rights, with the safety and well-being of patients.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT02698410/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02698410/SAP_001.pdf